CLINICAL TRIAL: NCT05541588
Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block For Postoperative Analgesia After Abdominal Hysterectomy; A Randomized Comparative Study
Brief Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block For Postoperative Analgesia After Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Khaled Abdou, clinical assistant professor -Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASUKH1
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB (Active Comparator): Erector Spinae Plane Block group
  Interventions: Procedure: peripheral nerve block
- QLB (Active Comparator): Quadratus Lumborum Block group
  Interventions: Procedure: peripheral nerve block

INTERVENTIONS:
Procedure: peripheral nerve block — ultrasound guided nerve block

SUMMARY:
The aim of this study is to compare the analgesic efficacy of erector spinae plane block and quadratus lumborum block after abdominal hysterectomy surgery and postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status 1-3.
* scheduled for abdominal hysterectomy surgery.

Exclusion Criteria:

* History of allergy to the medications used in the study.
* Contraindication to regional anesthesia as coagulopathy, local infection.
* Severe hepatic impairment (child C).
* Sever Renal dysfunction (creatinine clearance < 30).
* Psychiatric or mental disorder affecting patient ability to interpret VAS score.
* Body mass index (BMI) ≥ 40 or ≤ 18 kg/m2.
* ASA IV.
* Patient refusal.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females
Enrollment: 64 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 24 hours
  Post-operative pain severity assessed by visual analog scale (VAS) (range from 0-10., 0 no pain, 10 worst pain ).

SECONDARY OUTCOMES:
Cumulative post-operative opioid consumption | 24 hours
  opioid consumption
The onset of 1st analgesic request | 24 hours
  time needed for 1st request of rescue analgesia

OTHER OUTCOMES:
Incidence of complications | 24 hours
  postoperative nausea and vomiting(PONV), hematoma, local anaesthetic toxicity (LAT)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams univerisity, Cairo, Egypt